CLINICAL TRIAL: NCT04137913
Title: Project CHROMA (Cognitive Health Research on Musical Arts)
Brief Title: Cognitive Health Research on Musical Arts
Acronym: CHROMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-FY2019-355
Record Dates: First submitted 2019-10-08; First posted 2019-10-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Impairment; Creativity
Keywords: mild cognitive impairment; musical arts; whole brain network; cognition; aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Half the participants will be placed in the experimental group while the other half will be placed in the non wait-list control group (termed creative reading group to participants). Individuals in the control group will not be given the music intervention during their enrollment in the study. Due to the lack of funds, the research team is unable to provide individuals in the control group with the intervention after the study. Participants in the control group will be told that they have been placed in the creative reading group. They will receive a creativity book to read at the completion of their last visit. A post-study survey will be sent to the control group to minimize the possibility that control participants know that they're in the control group.
Masking Description: Due to limited funding, the research team is unable to conduct a truly randomized clinical trial. Research staff assessing baseline assessment (pre-intervention) and follow-up assessments (post-intervention) will not be intentionally masked. Participants also will not be masked. During the screening process, participants are told that they are randomized into a certain group: creative music and creative reading.They are informed which group they have been assigned to at their baseline visit because each group requires a different time commitment (music: requires coming in 3x a week for 6 weeks. reading/control: doesn't involve extra time commitment outside of the two research visits).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Individuals in the music group will complete two assessment visit (pre-intervention and post-intervention). After their baseline visit, they will participate in a 6-week group music class, scheduled for 2 hours a day, 3 days a week. The daily music workshops will be led by a musician associated with the Rice Shepherd School of Music. Each week will be carefully scaled in difficulty, with the workshops becoming progressively more sophisticated. For instance, the first week's listening will focus on short and more familiar works such as instrumental etudes and folk songs. Gradually, the instructor will build towards symphonic movements, as well as more unfamiliar and experimental music. The course will culminate in creating a final composition.
  Interventions: Behavioral: Musical arts intervention
- Non-music group (No Intervention): Individuals in the non-music group will complete two assessment visits separated by 2-3 months. They will be asked not to participate in any other music-related courses during the time they are enrolled in the study. At the end of participation, participants will be given resources to seek out music classes.

INTERVENTIONS:
Behavioral: Musical arts intervention — A 6-week group music class that incorporates listening, theory, performance, and creation of music.
  Arms: Music Group

SUMMARY:
This study is designed to assess the therapeutic effect that music creativity engagement has on cognition and social/emotional well-being, with a special interest in quantifying the associated connectivity changes in the brain. Investigators will measure the effect that a creative music intervention has on health-related outcomes for mild cognitive impairment (MCI) patients using novel neural markers, laboratory-based cognitive tasks, assessments of loneliness, perceptions of stress, and social support.

DETAILED DESCRIPTION:
4.1 Design A six-week creative music course designed by Dr. Brandt and the other award-winning composers of Musiqa will be taught by graduate student composers from the Rice Shepherd School of Music. To make the course as accessible as possible, participants will not need to be able to read musical notation or have any prior musical background, and we will utilize established ways of effactively inspiring untrained musicians (26). It will meet 4 hours per day, for five days a week. The daily music workshops will have four components: listening, theory, performance, and creation (Table 1). Each week will be carefully scaled in difficulty, with the workshops becoming progressively more sophisticated.

4.2 Study Setting The study may take place at different locations depending on assessments. Screening assessments will take place over the phone with a research staff member. Interested individuals will complete the first visit for a baseline blood draw, health assessments, cognitive tasks, and social and emotional well-being assessments at Rice University's BioScience Research Collaborative (BRC) building, Suite 140. Participants will be brought to the BRC building by their caregiver or family member. Baseline neuroimaging will be performed at Houston Methodist Research Institute Translational Imaging Center. Participants will be randomly assigned to either the experimental group (music group) or the control group (non-music group).

Participants in the experimental group will undergo a 6-week music training headed by a musician associated with the Rice's Shepherd School of Music. The music intervention will take place on the main campus of Rice University or at the Bioscience Research Collaborative, Rm 707.

Additionally, the social, physical, and emotional wellbeing of the participant and the caregiver (if present) will be assessed with a battery of questionnaires before and after the intervention.

4.3 Recruitment and Data Collection Procedures

Participant Recruitment:

Recruitment. Participants with mild cognitive impairment will be recruited from medical centers, such as Baylor College of Medicine and UT Health. We have partnered with Dr. Jennifer M. Stinson at the Alzheimer's Disease and Memory Disorders Center of BCM, a leading research and clinical center that manages the diagnosis and treatment of more than 3,000 MCI patients a year, along with providing them with avenues for participation in clinical trials. We will establish partnerships with medical facilities that treat mild cognitive impaired patients in order to advertise our study. Specifically, we will obtain IRB approval from outside institutions (e.g., UT Health McGovern Medical School, Baylor St. Luke's, Houston Methodist Hospital, and Baylor College of Medicine) in order to recruit participants directly from medical clinics. Upon approval, physicians may provide us access to their patient clinic schedule, access to patient portal (e.g. EPOCH at Baylor College of Medicine), or the ability to receive patient referrals from the treating physician. Furthermore, this study will be listed on Trial Match, a clinical studies matching service provided by Alzheimer's Association, and on ResearchMatch, a free and secure online tool created by academic institutions across the country.

In addition, we will recruit older adult subjects without MCI by proactively posting and distributing flyers at retirement homes, assisted-living homes, community centers, medical facilities, neighborhoods, and community events. These flyers will contain details about our study as well as an email and phone number for further contact. We will also advertise our study on newspapers, social media groups, and/or radio/television.

Screening. Participants will be screened over the phone or via online screening form to ensure that they meet general criteria for study participation. If we sense during the phone or online screening that a participant displays cognitive deficits that could not be definitively confirmed, we will send him or her a copy of the consent form. If the participant does not exhibit noticeable cognitive deficits during the phone screening stage, these three questions will be asked when they come in for their first visit, prior to signing the consent form. After the participant reads the consent form, the participant will be asked if they have any questions or need further explanation of what is being asked of them. We will ask three questions to confirm that the participant shows acceptable understanding of his/her participation in the study. These questions seek to verify that the participant understands what involvement in the study entails and his/her ability to refuse participation at any point of the study. If they are able to explain the above, they are considered cognitively competent to participate in the study.

For participants with MCI, formal confirmation from the medical doctor is needed to confirm medical diagnosis of mild cognitive impairment. Thus, eligible individuals will be sent an online version or hardcopy version of a medical release form that will be signed and mailed to both us and the doctor. MCI diagnosis is not required for participation but those who claim to have MCI must provide medical documents to confirm this diagnosis.

Design and Key Protocol Components:

Participants will be instructed to adhere to the regimented breakfast the morning of baseline and follow-up assessment visits. We recognize that this variation may alter internal validity; however, it will maintain external validity (studies have demonstrated that this level of variation has a modest impact on inflammation (27). Participants will also be asked to avoid any strenuous physical activity for 48 hours before the baseline and follow-up assessment visits. All visits will be audio recorded for quality control purposes and surveillance purposes.

As mentioned earlier, baseline and follow-up visits will take place at the BRC building on Main street and Houston Methodist Research Institute Translational Imaging Center for both experimental (music group) and control (non-music group) groups. Visits will be scheduled to start between 7:30 AM and 10:30 AM.

Participants in the musical group will participate in a 6-week group music course (3 days a week, 2 hours per day) after their baseline visit. Follow-up assessments for the musical group will occur within 2-4 weeks of completion of the 6-week music course. Caregivers will be given the option of mingling with the other caregivers or have relief from care.

Participants in the creative reading group (control group) will be asked not to participate in any music-related activities between their baseline and follow-up visits. Baseline and follow-up visits will be scheduled within 3-4 months of each other or mirror the approximate time gap between the baseline visit and follow-up visit for a participant in the music group (experimental group). Those who were not selected for the music course will be given a book with a short survey 1-3 weeks after the follow-up (final) in-person visit.

Participant Contact before Baseline and Follow-up Visits:

Before the baseline and follow-up assessment visits, a research staff member will call participants (1 day prior) and remind them of the visit. Given that inflammatory markers may be elevated during acute illnesses, such as upper respiratory infections, we will ask them if they are experiencing any illness symptoms (e.g., fever, congestion, sore throat, or acute infections due to injury). During this phone call, we will also ask and ensure they have followed directions not to exercise for 48 hours prior to the visit, to adhere to the regimented breakfast list, and to avoid wearing metal objects. Participants will be rescheduled for a different time if they are ill or did not follow the exercise restriction.

Assessments:

After the participant reads the consent form, the participant will be asked if they have any questions or need further explanation of what is being asked of them. We will ask three questions to confirm that the participant shows acceptable understanding of participation for eligibility. Study personnel will ensure comprehension by asking what tasks are expected of them with their participation and ask them to explain what they would do if they decided they no longer want to participate in the study. If they are able to adequately answer the above questions, they are considered cognitively competent to participate in the study.

Baseline and follow-up assessments will take place on campus at the Bioscience Research Collaborative (BRC) in suite 140 and at the Houston Methodist Research Institute Translational Imaging Center. Visits will be scheduled to start between 7:30 AM and 10:30 AM. A research coordinator will provide a detailed description of the study, answer questions, and obtain written informed consent. Participants will complete questionnaires, cognitive tasks, and health assessments (e.g., measuring heart rate, weight, blood pressure, and waistline measurements) and have blood drawn. Caregivers, if consented to participate, will fill out self-report questionnaires pertaining to social and emotional well-being. Neural activity using the fMRI will be collected in the Houston Methodist Research Institute Translational Imaging Center. After completing the music course, participants will be scheduled for one follow-up visit. The baseline and follow-up visits should last about 3.5-4.5 hours at the BRC and about 1.5 hours at Houston Methodist Research Institute Translational Imaging Center.

Financial Compensation:

Participants with mild cognitive impairment will be reimbursed at baseline and follow-up visits. For each visit, MCI participants will be compensated $50, for a total of $100 by the end of the study. Completion of the EEfRT task amd Monetary Incentive Delay (MID) task will result in an addition of $5-20 at the baseline visit (based on performance of the task). Participants will be provided with parking validations for each assessment visit and during the 6-week music course.

ELIGIBILITY:
Inclusion Criteria for participants:

1. Over the age of 70, unless diagnosed with early to moderate mild cognitive impairment (self-described and confirmed by physician).
2. Able to read and write in English
3. Cognitively competent to participate (i.e. correctly answers three questions to confirm comprehension of participation)
4. Demonstrate ability to follow instructions

Exclusion Criteria for participants:

1. Below the age of 70 and not diagnosed with MCI.
2. Significant visual or auditory impairment resulting in the inability to read and/or hear the questionnaires
3. Class III heart failure
4. Autoimmune and/or inflammatory disorders
5. Any implanted medical device that renders one unable to undergo fMRI scanning
6. Pregnant or nursing women
7. Weight > 300lb or BMI over 40
8. Professional musician
9. Comorbid diagnosis of Parkinson's Disease
10. Dental implants or extensive dental work that impedes collection of good-quality fMRI data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional resting state brain activity at follow-up visit. | Functional magnetic resonance imaging will be obtained at enrollment and within one month since the completion of the music course.
  Modularity and flexibility will act as quantifiers of neural activity. Modularity is the degree to which neural activity within a group of brain regions is more highly correlated than is activity between such groups, and flexibility is the dynamic reorganization of these groups.
Mean change from baseline in level of creativity using scores on Guilford's alternative Uses Divergent Thinking Test | Creativity will be measured at enrollment and within one month since the completion of the music course.
  Total scores are derived based on fluency, flexibility, originality, and elaboration. Higher scores indicate greater creativity. There is no max score.
Mean change in scores from baseline in perceived social support subscales of the Medical Outcomes Studies, including emotional support, tangible support, affectionate support, and positive social interactions. | Creativity will be measured at enrollment and within one month since the completion of the music course.
  Scores are transformed to a 0-100 scale. Higher scores on the self-report social support scale indicate a larger degree of perceived social support in each of these domains: emotional support, tangible support, affectionate support, and positive social interaction.
Mean change from baseline in quality of life scores each subscale of the SF-36 | Quality of life will be measured at enrollment and within one month since the completion of the music course.
  Eight subscales measuring quality of life are scored out of 100. These subscales include: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general and health. Lower scores indicate greater disability.
Mean change from baseline in inhibition and inhibition/switching trials on the color-word interference test of the Delis Kaplan Executive Function System (DKEFS) | Cognitive scores will be measured at enrollment and within one month since the completion of the music course.
  Higher scores for inhibition and inhibition/switching trials indicate greater executive functioning. Scaled and raw scores will be assessed. There is no minimum and maximum score.
Mean change from baseline in cognitive scores (digit span forward, digit span backward, digit span sequencing, and total raw score) on the digit span test of the Wechsler Adult Intelligence Scale (WAIS). | Cognitive scores will be measured at enrollment and within one month since the completion of the music course.
  Higher scores indicate greater working memory ability. Each subscale (forward, backward, and sequencing) has a maximum score of 16. The maximum total raw score is 48.
Mean change from baseline in perseverative errors on the Wisconsin Card Sorting Test (WCST) | Cognitive scores will be measured at enrollment and within one month since the completion of the music course.
  The Wisconsin Card Sorting Test assess executive control. Scores on the WCST are based on percentages of categories achieved, errors, and perseveration errors. Greater number of perseverative errors indicate poorer executive control.
Mean change from baseline in affect scores on the Positive and Negative Affect Scale | Daily affect scores will be measured for 7 days after enrollment and 7 days after the final follow-up visit that will take place within 1 month after the completion of the music course.
  Two scales measuring positive and negative affect. Scores range from 10-50 on each scale. Higher scores on positive affect scale indicate higher levels of positive affect. Lower scores on the negative affect scale indicate lower levels of negative affect.
Mean change from baseline in emotion regulation scores on the Emotional Regulation Scale | Emotion regulation scores will be measured at enrollment and at the follow-up visit that will take place within one month after the completion of the music course.
  The self-report questionnaire measures the extent to which one uses cognitive appraisal or suppression techniques to regulate emotions. Higher scores on each subscale indicate greater use of that regulation strategy. Scores are continuous. The emotional reappraisal scale has a max score of 42. The emotional suppression scale has a max score of 28.

SECONDARY OUTCOMES:
Mean change in inflammation from enrollment (baseline) to follow-up visit | Blood will be drawn at enrollment and within one month after the completion of the music study (for experimental group).
  Serum cytokines and C-reactive protein will be assessed as a biomarker of systemic inflammation. These specific cytokines include: T-cell stimulated IL-6, TNFa, IFNg, IL17a, IL-2. Higher volume (pg/mL) of these individual proinflammatory biomarkers indicates higher levels of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Fagundes, Ph.D., Principal Investigator — William Marsh Rice University
Locations (1):
- Rice University Bioscience Research Collaborative, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karmonik C, Brandt A, Anderson J, Brooks F, Lytle J, Silverman E, Frazier JT. Music Listening modulates Functional Connectivity and Information Flow in the Human Brain. Brain Connect. 2016 Oct;6(8):632-641. doi: 10.1089/brain.2016.0428. Epub 2016 Jul 27. PMID 27464741
- [Background] Yue Q, Martin RC, Fischer-Baum S, Ramos-Nunez AI, Ye F, Deem MW. Brain Modularity Mediates the Relation between Task Complexity and Performance. J Cogn Neurosci. 2017 Sep;29(9):1532-1546. doi: 10.1162/jocn_a_01142. Epub 2017 May 4. PMID 28471728
- [Background] Jaremka LM, Andridge RR, Fagundes CP, Alfano CM, Povoski SP, Lipari AM, Agnese DM, Arnold MW, Farrar WB, Yee LD, Carson WE 3rd, Bekaii-Saab T, Martin EW Jr, Schmidt CR, Kiecolt-Glaser JK. Pain, depression, and fatigue: loneliness as a longitudinal risk factor. Health Psychol. 2014 Sep;33(9):948-57. doi: 10.1037/a0034012. Epub 2013 Aug 19. PMID 23957903
- [Background] Brandt A, Gebrian M, Slevc LR. Music and early language acquisition. Front Psychol. 2012 Sep 11;3:327. doi: 10.3389/fpsyg.2012.00327. eCollection 2012. PMID 22973254
- [Background] Parbery-Clark A, Skoe E, Lam C, Kraus N. Musician enhancement for speech-in-noise. Ear Hear. 2009 Dec;30(6):653-61. doi: 10.1097/AUD.0b013e3181b412e9. PMID 19734788
- [Background] Kraus N, Slater J, Thompson EC, Hornickel J, Strait DL, Nicol T, White-Schwoch T. Music enrichment programs improve the neural encoding of speech in at-risk children. J Neurosci. 2014 Sep 3;34(36):11913-8. doi: 10.1523/JNEUROSCI.1881-14.2014. PMID 25186739
- [Background] Bengtsson SL, Csikszentmihalyi M, Ullen F. Cortical regions involved in the generation of musical structures during improvisation in pianists. J Cogn Neurosci. 2007 May;19(5):830-42. doi: 10.1162/jocn.2007.19.5.830. PMID 17488207
- [Background] Limb CJ, Braun AR. Neural substrates of spontaneous musical performance: an FMRI study of jazz improvisation. PLoS One. 2008 Feb 27;3(2):e1679. doi: 10.1371/journal.pone.0001679. PMID 18301756
- [Background] He J, Sun J, Deem MW. Spontaneous emergence of modularity in a model of evolving individuals and in real networks. Phys Rev E Stat Nonlin Soft Matter Phys. 2009 Mar;79(3 Pt 1):031907. doi: 10.1103/PhysRevE.79.031907. Epub 2009 Mar 17. PMID 19391971
- [Background] Park JM, Niestemski LR, Deem MW. Quasispecies theory for evolution of modularity. Phys Rev E Stat Nonlin Soft Matter Phys. 2015 Jan;91(1):012714. doi: 10.1103/PhysRevE.91.012714. Epub 2015 Jan 28. PMID 25679649
- [Background] Holmen K, Ericsson K, Winblad B. Social and emotional loneliness among non-demented and demented elderly people. Arch Gerontol Geriatr. 2000 Dec;31(3):177-192. doi: 10.1016/s0167-4943(00)00070-4. PMID 11154772
- [Background] Steptoe A, Shankar A, Demakakos P, Wardle J. Social isolation, loneliness, and all-cause mortality in older men and women. Proc Natl Acad Sci U S A. 2013 Apr 9;110(15):5797-801. doi: 10.1073/pnas.1219686110. Epub 2013 Mar 25. PMID 23530191
- [Background] Stuckey HL, Nobel J. The connection between art, healing, and public health: a review of current literature. Am J Public Health. 2010 Feb;100(2):254-63. doi: 10.2105/AJPH.2008.156497. Epub 2009 Dec 17. PMID 20019311
- [Background] Jaremka LM, Fagundes CP, Glaser R, Bennett JM, Malarkey WB, Kiecolt-Glaser JK. Loneliness predicts pain, depression, and fatigue: understanding the role of immune dysregulation. Psychoneuroendocrinology. 2013 Aug;38(8):1310-7. doi: 10.1016/j.psyneuen.2012.11.016. Epub 2012 Dec 27. PMID 23273678
- [Background] Chen M, Deem MW. Development of modularity in the neural activity of children's brains. Phys Biol. 2015 Jan 26;12(1):016009. doi: 10.1088/1478-3975/12/1/016009. PMID 25619207
- [Background] Fagundes CP, Lindgren ME, Shapiro CL, Kiecolt-Glaser JK. Child maltreatment and breast cancer survivors: social support makes a difference for quality of life, fatigue and cancer stress. Eur J Cancer. 2012 Mar;48(5):728-36. doi: 10.1016/j.ejca.2011.06.022. PMID 21752636
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Raglio A, Attardo L, Gontero G, Rollino S, Groppo E, Granieri E. Effects of music and music therapy on mood in neurological patients. World J Psychiatry. 2015 Mar 22;5(1):68-78. doi: 10.5498/wjp.v5.i1.68. PMID 25815256
- [Background] Ramos-Nunez AI, Fischer-Baum S, Martin RC, Yue Q, Ye F, Deem MW. Static and Dynamic Measures of Human Brain Connectivity Predict Complementary Aspects of Human Cognitive Performance. Front Hum Neurosci. 2017 Aug 24;11:420. doi: 10.3389/fnhum.2017.00420. eCollection 2017. PMID 28883789
- [Background] Newman ME. Modularity and community structure in networks. Proc Natl Acad Sci U S A. 2006 Jun 6;103(23):8577-82. doi: 10.1073/pnas.0601602103. Epub 2006 May 24. PMID 16723398
- [Background] Galland L. Diet and inflammation. Nutr Clin Pract. 2010 Dec;25(6):634-40. doi: 10.1177/0884533610385703. PMID 21139128
- [Background] Breuer FA, Blaimer M, Heidemann RM, Mueller MF, Griswold MA, Jakob PM. Controlled aliasing in parallel imaging results in higher acceleration (CAIPIRINHA) for multi-slice imaging. Magn Reson Med. 2005 Mar;53(3):684-91. doi: 10.1002/mrm.20401. PMID 15723404
- [Background] Knutson B, Bhanji JP, Cooney RE, Atlas LY, Gotlib IH. Neural responses to monetary incentives in major depression. Biol Psychiatry. 2008 Apr 1;63(7):686-92. doi: 10.1016/j.biopsych.2007.07.023. Epub 2007 Oct 4. PMID 17916330
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Eysenck HJ, Furnham A. Personality and the Barron-Welsh Art Scale. Percept Mot Skills. 1993 Jun;76(3 Pt 1):837-8. doi: 10.2466/pms.1993.76.3.837. PMID 8321595
- [Background] Baum A, Cohen L, Hall M. Control and intrusive memories as possible determinants of chronic stress. Psychosom Med. 1993 May-Jun;55(3):274-86. doi: 10.1097/00006842-199305000-00005. PMID 8346335
- [Background] BARRON F. The disposition toward originality. J Abnorm Psychol. 1955 Nov;51(3):478-85. doi: 10.1037/h0048073. No abstract available. PMID 13285986
- [Background] Treadway MT, Buckholtz JW, Schwartzman AN, Lambert WE, Zald DH. Worth the 'EEfRT'? The effort expenditure for rewards task as an objective measure of motivation and anhedonia. PLoS One. 2009 Aug 12;4(8):e6598. doi: 10.1371/journal.pone.0006598. PMID 19672310
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Seeman TE, Berkman LF. Structural characteristics of social networks and their relationship with social support in the elderly: who provides support. Soc Sci Med. 1988;26(7):737-49. doi: 10.1016/0277-9536(88)90065-2. PMID 3358145
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Background] Ingram SS, Seo PH, Martell RE, Clipp EC, Doyle ME, Montana GS, Cohen HJ. Comprehensive assessment of the elderly cancer patient: the feasibility of self-report methodology. J Clin Oncol. 2002 Feb 1;20(3):770-5. doi: 10.1200/JCO.2002.20.3.770. PMID 11821460
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Demark-Wahnefried W, Clipp EC, McBride C, Lobach DF, Lipkus I, Peterson B, Clutter Snyder D, Sloane R, Arbanas J, Kraus WE. Design of FRESH START: a randomized trial of exercise and diet among cancer survivors. Med Sci Sports Exerc. 2003 Mar;35(3):415-24. doi: 10.1249/01.MSS.0000053704.28156.0F. PMID 12618570
- [Background] Blair SN, Haskell WL, Ho P, Paffenbarger RS Jr, Vranizan KM, Farquhar JW, Wood PD. Assessment of habitual physical activity by a seven-day recall in a community survey and controlled experiments. Am J Epidemiol. 1985 Nov;122(5):794-804. doi: 10.1093/oxfordjournals.aje.a114163. PMID 3876763
- [Background] Taylor CB, Coffey T, Berra K, Iaffaldano R, Casey K, Haskell WL. Seven-day activity and self-report compared to a direct measure of physical activity. Am J Epidemiol. 1984 Dec;120(6):818-24. doi: 10.1093/oxfordjournals.aje.a113954. PMID 6507425
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Bower JE, Ganz PA, Desmond KA, Bernaards C, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer. 2006 Feb 15;106(4):751-8. doi: 10.1002/cncr.21671. PMID 16400678
- [Background] Collado-Hidalgo A, Bower JE, Ganz PA, Cole SW, Irwin MR. Inflammatory biomarkers for persistent fatigue in breast cancer survivors. Clin Cancer Res. 2006 May 1;12(9):2759-66. doi: 10.1158/1078-0432.CCR-05-2398. PMID 16675568
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Hartrick CT, Kovan JP, Shapiro S. The numeric rating scale for clinical pain measurement: a ratio measure? Pain Pract. 2003 Dec;3(4):310-6. doi: 10.1111/j.1530-7085.2003.03034.x. PMID 17166126
- [Background] Miro J, Castarlenas E, Huguet A. Evidence for the use of a numerical rating scale to assess the intensity of pediatric pain. Eur J Pain. 2009 Nov;13(10):1089-95. doi: 10.1016/j.ejpain.2009.07.002. Epub 2009 Sep 1. PMID 19726211
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Potts MK, Daniels M, Burnam MA, Wells KB. A structured interview version of the Hamilton Depression Rating Scale: evidence of reliability and versatility of administration. J Psychiatr Res. 1990;24(4):335-50. doi: 10.1016/0022-3956(90)90005-b. PMID 2090831
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cohen S, Tyrrell DA, Smith AP. Psychological stress and susceptibility to the common cold. N Engl J Med. 1991 Aug 29;325(9):606-12. doi: 10.1056/NEJM199108293250903. PMID 1713648
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Berney LR, Blane DB. Collecting retrospective data: accuracy of recall after 50 years judged against historical records. Soc Sci Med. 1997 Nov;45(10):1519-25. doi: 10.1016/s0277-9536(97)00088-9. PMID 9351141
- [Background] Pugh H, Power C, Goldblatt P, Arber S. Women's lung cancer mortality, socio-economic status and changing smoking patterns. Soc Sci Med. 1991;32(10):1105-10. doi: 10.1016/0277-9536(91)90086-r. PMID 2068593
- [Background] Bower JE. Behavioral symptoms in patients with breast cancer and survivors. J Clin Oncol. 2008 Feb 10;26(5):768-77. doi: 10.1200/JCO.2007.14.3248. PMID 18258985
- [Background] Bower JE, Ganz PA, Aziz N, Fahey JL, Cole SW. T-cell homeostasis in breast cancer survivors with persistent fatigue. J Natl Cancer Inst. 2003 Aug 6;95(15):1165-8. doi: 10.1093/jnci/djg0019. PMID 12902446
- [Background] Bower JE, Ganz PA, Aziz N. Altered cortisol response to psychologic stress in breast cancer survivors with persistent fatigue. Psychosom Med. 2005 Mar-Apr;67(2):277-80. doi: 10.1097/01.psy.0000155666.55034.c6. PMID 15784794
- [Background] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Background] Donovan KA, Small BJ, Andrykowski MA, Munster P, Jacobsen PB. Utility of a cognitive-behavioral model to predict fatigue following breast cancer treatment. Health Psychol. 2007 Jul;26(4):464-72. doi: 10.1037/0278-6133.26.4.464. PMID 17605566
- [Background] Fagundes CP, Murray DM, Hwang BS, Gouin JP, Thayer JF, Sollers JJ 3rd, Shapiro CL, Malarkey WB, Kiecolt-Glaser JK. Sympathetic and parasympathetic activity in cancer-related fatigue: more evidence for a physiological substrate in cancer survivors. Psychoneuroendocrinology. 2011 Sep;36(8):1137-47. doi: 10.1016/j.psyneuen.2011.02.005. Epub 2011 Mar 9. PMID 21388744
- [Background] Bower JE, Ganz PA, Aziz N, Fahey JL. Fatigue and proinflammatory cytokine activity in breast cancer survivors. Psychosom Med. 2002 Jul-Aug;64(4):604-11. doi: 10.1097/00006842-200207000-00010. PMID 12140350
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Maes M, Song C, Lin A, De Jongh R, Van Gastel A, Kenis G, Bosmans E, De Meester I, Benoy I, Neels H, Demedts P, Janca A, Scharpe S, Smith RS. The effects of psychological stress on humans: increased production of pro-inflammatory cytokines and a Th1-like response in stress-induced anxiety. Cytokine. 1998 Apr;10(4):313-8. doi: 10.1006/cyto.1997.0290. PMID 9617578
- [Background] Lutgendorf SK, Garand L, Buckwalter KC, Reimer TT, Hong SY, Lubaroff DM. Life stress, mood disturbance, and elevated interleukin-6 in healthy older women. J Gerontol A Biol Sci Med Sci. 1999 Sep;54(9):M434-9. doi: 10.1093/gerona/54.9.m434. PMID 10536645
- [Background] DeRijk R, Michelson D, Karp B, Petrides J, Galliven E, Deuster P, Paciotti G, Gold PW, Sternberg EM. Exercise and circadian rhythm-induced variations in plasma cortisol differentially regulate interleukin-1 beta (IL-1 beta), IL-6, and tumor necrosis factor-alpha (TNF alpha) production in humans: high sensitivity of TNF alpha and resistance of IL-6. J Clin Endocrinol Metab. 1997 Jul;82(7):2182-91. doi: 10.1210/jcem.82.7.4041. PMID 9215292
- [Background] Zhou D, Kusnecov AW, Shurin MR, DePaoli M, Rabin BS. Exposure to physical and psychological stressors elevates plasma interleukin 6: relationship to the activation of hypothalamic-pituitary-adrenal axis. Endocrinology. 1993 Dec;133(6):2523-30. doi: 10.1210/endo.133.6.8243274.
- [Background] Lutgendorf SK, Logan H, Costanzo E, Lubaroff D. Effects of acute stress, relaxation, and a neurogenic inflammatory stimulus on interleukin-6 in humans. Brain Behav Immun. 2004 Jan;18(1):55-64. doi: 10.1016/s0889-1591(03)00090-4. PMID 14651947
- [Background] Brydon L, Edwards S, Mohamed-Ali V, Steptoe A. Socioeconomic status and stress-induced increases in interleukin-6. Brain Behav Immun. 2004 May;18(3):281-90. doi: 10.1016/j.bbi.2003.09.011. PMID 15050655
- [Background] Segerstrom SC, Miller GE. Psychological stress and the human immune system: a meta-analytic study of 30 years of inquiry. Psychol Bull. 2004 Jul;130(4):601-30. doi: 10.1037/0033-2909.130.4.601. PMID 15250815
- [Background] Kiecolt-Glaser JK, Preacher KJ, MacCallum RC, Atkinson C, Malarkey WB, Glaser R. Chronic stress and age-related increases in the proinflammatory cytokine IL-6. Proc Natl Acad Sci U S A. 2003 Jul 22;100(15):9090-5. doi: 10.1073/pnas.1531903100. Epub 2003 Jul 2. PMID 12840146
- [Background] Dentino AN, Pieper CF, Rao MK, Currie MS, Harris T, Blazer DG, Cohen HJ. Association of interleukin-6 and other biologic variables with depression in older people living in the community. J Am Geriatr Soc. 1999 Jan;47(1):6-11. doi: 10.1111/j.1532-5415.1999.tb01894.x. PMID 9920223
- [Background] Maes M, Lin AH, Delmeire L, Van Gastel A, Kenis G, De Jongh R, Bosmans E. Elevated serum interleukin-6 (IL-6) and IL-6 receptor concentrations in posttraumatic stress disorder following accidental man-made traumatic events. Biol Psychiatry. 1999 Apr 1;45(7):833-9. doi: 10.1016/s0006-3223(98)00131-0. PMID 10202570
- [Background] Glaser R, Robles TF, Sheridan J, Malarkey WB, Kiecolt-Glaser JK. Mild depressive symptoms are associated with amplified and prolonged inflammatory responses after influenza virus vaccination in older adults. Arch Gen Psychiatry. 2003 Oct;60(10):1009-14. doi: 10.1001/archpsyc.60.10.1009. PMID 14557146
- [Background] Suarez EC, Lewis JG, Krishnan RR, Young KH. Enhanced expression of cytokines and chemokines by blood monocytes to in vitro lipopolysaccharide stimulation are associated with hostility and severity of depressive symptoms in healthy women. Psychoneuroendocrinology. 2004 Oct;29(9):1119-28. doi: 10.1016/j.psyneuen.2004.01.002. PMID 15219635
- [Background] Pitsavos C, Panagiotakos DB, Papageorgiou C, Tsetsekou E, Soldatos C, Stefanadis C. Anxiety in relation to inflammation and coagulation markers, among healthy adults: the ATTICA study. Atherosclerosis. 2006 Apr;185(2):320-6. doi: 10.1016/j.atherosclerosis.2005.06.001. Epub 2005 Jul 11. PMID 16005881
- [Background] Marx J. Cancer research. Inflammation and cancer: the link grows stronger. Science. 2004 Nov 5;306(5698):966-8. doi: 10.1126/science.306.5698.966. No abstract available. PMID 15528423
- [Background] Ershler WB, Keller ET. Age-associated increased interleukin-6 gene expression, late-life diseases, and frailty. Annu Rev Med. 2000;51:245-70. doi: 10.1146/annurev.med.51.1.245. PMID 10774463
- [Background] Pradhan AD, Manson JE, Rifai N, Buring JE, Ridker PM. C-reactive protein, interleukin 6, and risk of developing type 2 diabetes mellitus. JAMA. 2001 Jul 18;286(3):327-34. doi: 10.1001/jama.286.3.327. PMID 11466099
- [Background] Musselman DL, Miller AH, Porter MR, Manatunga A, Gao F, Penna S, Pearce BD, Landry J, Glover S, McDaniel JS, Nemeroff CB. Higher than normal plasma interleukin-6 concentrations in cancer patients with depression: preliminary findings. Am J Psychiatry. 2001 Aug;158(8):1252-7. doi: 10.1176/appi.ajp.158.8.1252. PMID 11481159
- [Background] Miller AH. Neuroendocrine and immune system interactions in stress and depression. Psychiatr Clin North Am. 1998 Jun;21(2):443-63. doi: 10.1016/s0193-953x(05)70015-0. PMID 9670236
- [Background] Maes M, Bosmans E, De Jongh R, Kenis G, Vandoolaeghe E, Neels H. Increased serum IL-6 and IL-1 receptor antagonist concentrations in major depression and treatment resistant depression. Cytokine. 1997 Nov;9(11):853-8. doi: 10.1006/cyto.1997.0238. PMID 9367546
- [Background] Irwin M. Psychoneuroimmunology of depression: clinical implications. Brain Behav Immun. 2002 Feb;16(1):1-16. doi: 10.1006/brbi.2001.0654. PMID 11846437
- [Background] Zorrilla EP, Luborsky L, McKay JR, Rosenthal R, Houldin A, Tax A, McCorkle R, Seligman DA, Schmidt K. The relationship of depression and stressors to immunological assays: a meta-analytic review. Brain Behav Immun. 2001 Sep;15(3):199-226. doi: 10.1006/brbi.2000.0597. PMID 11566046
- [Background] Irwin MR, Wang M, Campomayor CO, Collado-Hidalgo A, Cole S. Sleep deprivation and activation of morning levels of cellular and genomic markers of inflammation. Arch Intern Med. 2006 Sep 18;166(16):1756-62. doi: 10.1001/archinte.166.16.1756. PMID 16983055
- [Background] Korenromp IH, Grutters JC, van den Bosch JM, Zanen P, Kavelaars A, Heijnen CJ. Reduced Th2 cytokine production by sarcoidosis patients in clinical remission with chronic fatigue. Brain Behav Immun. 2011 Oct;25(7):1498-502. doi: 10.1016/j.bbi.2011.06.004. Epub 2011 Jun 13. PMID 21693184
- [Background] Fagundes CP, Glaser R, Alfano CM, Bennett JM, Povoski SP, Lipari AM, Agnese DM, Yee LD, Carson WE 3rd, Farrar WB, Malarkey WB, Kiecolt-Glaser JK. Fatigue and herpesvirus latency in women newly diagnosed with breast cancer. Brain Behav Immun. 2012 Mar;26(3):394-400. doi: 10.1016/j.bbi.2011.09.014. Epub 2011 Oct 2. PMID 21988771
- [Background] Schultze-Florey CR, Martinez-Maza O, Magpantay L, Breen EC, Irwin MR, Gundel H, O'Connor MF. When grief makes you sick: bereavement induced systemic inflammation is a question of genotype. Brain Behav Immun. 2012 Oct;26(7):1066-71. doi: 10.1016/j.bbi.2012.06.009. Epub 2012 Jun 23. PMID 22735772
- [Background] van Zuiden M, Heijnen CJ, van de Schoot R, Amarouchi K, Maas M, Vermetten E, Geuze E, Kavelaars A. Cytokine production by leukocytes of military personnel with depressive symptoms after deployment to a combat-zone: a prospective, longitudinal study. PLoS One. 2011;6(12):e29142. doi: 10.1371/journal.pone.0029142. Epub 2011 Dec 14. PMID 22195009
- [Background] Schwarz AJ, Gozzi A, Bifone A. Community structure and modularity in networks of correlated brain activity. Magn Reson Imaging. 2008 Sep;26(7):914-20. doi: 10.1016/j.mri.2008.01.048. Epub 2008 May 13. PMID 18479871
- [Background] Hattori H, Hattori C, Hokao C, Mizushima K, Mase T. Controlled study on the cognitive and psychological effect of coloring and drawing in mild Alzheimer's disease patients. Geriatr Gerontol Int. 2011 Oct;11(4):431-7. doi: 10.1111/j.1447-0594.2011.00698.x. Epub 2011 Apr 26. PMID 21518170
- [Background] Schafer JL, Graham JW. Missing data: our view of the state of the art. Psychol Methods. 2002 Jun;7(2):147-77. PMID 12090408
- [Background] Bonomo ME, Karmonik C, Brandt AK, Frazier JT. Correlations between whole-brain modularity and flexibility distinguish music and speech perception. (submitted).
- [Background] Kachanathu SJ, Bhatia P, Nuhmani S, Vennu V. Efficacy of music listening with conventional physiotherapy management on sub-acute stroke patients. 2013;7.
- [Background] Deem MW. Statistical Mechanics of Modularity and Horizontal Gene Transfer. Annu Rev Condens Matter Phys. 2013;4(1):287-311.
- [Background] The Arts and Aging: Building the Science. National Endowment for the Arts Office of Research and Analysis; 2013.
- [Background] Hickey M. Music Outside the Lines: Ideas for Composing K-12 Music Classrooms. Oxford: Oxford University Press; 2012. 192 p.
- [Background] Wechsler D. WAIS-IV. In: Wechsler Adult Intelligence. San Antonio, Texas: NCS Pearson; 2008. p. 1-3.
- [Background] Delis DC, Kaplan E, Kramer J. Delis-Kaplan Executive Function System. Psychological Corporation; 2001.
- [Background] Heaton RK, Chelune GJ, Talley J.L. Wisconsin Card Sorting Test manual. Odessa, Florida: Psychological ASsessment Resources, Inc; 1993.
- [Background] Guilford JP. The nature of human intelligence. New York: McGraw-Hill; 1967.
- [Background] Rosen JC. The Barron-Welsh Art Scale as a predictor of originality and level of ability among artists. J Appl Psychol. 1956;39(5):366.
- [Background] Welsh GS, Gough HB, Hall WB, Bradley P. Barron Welsh Art Scale. Mind Garden; 1987. 84 p.
- [Background] Rammstedt B, John OP. Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. J Res Personal. 2007 Feb 1;41(1):203-12.
- [Background] Berkman LF, Kawachi I. Social Epidemiology. Oxford University Press; 2000. 414 p.
- [Background] Deci EL, Ryan RM. The "What" and "Why" of Goal Pursuits: Human Needs and the Self-Determination of Behavior. Psychol Inq. 2000 Oct;11(4):227-68.
- [Background] Jacobsen P, Donovan K. Cancer and fatigue: Insights from studies of women treated for breast cancer. In: Fatigue as a window to the brain. Cambridge, Massachusetts: MIT Press; 2005. p. 265-80.
- [Background] McCaffery M, Beebe A. Pain: Clinical manual for nursing practice. St. Louis, MO: Mosby; 1989.
- [Background] Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. Appl Psychol Meas. 1977 Jun 1;1(3):385-401.
- [Background] Basco MR, Krebaum SR, Rush AJ. Outcome measures of depression. In: Strupp HH, Horowitz LM, Lambert MJ, editors. Measuring Patient Changes in Mood, Anxiety, and Personality disorders. Washington D. C.: American Psychological Association; 1997. p. 207-45.
- [Background] Shahid A, Wilkinson K, Marcu S, Shapiro CM, editors. Hamilton Rating Scale for Depression. In: STOP, THAT and One Hundred Other Sleep Scales [Internet]. New York: Springer-Verlag; 2012 [cited 2019 May 14]. p. 187-90. Available from: https://www.springer.com/us/book/9781441998927
- [Background] Henderson AG, Byrne DG, Duncan-Jones P. Neurosis and the social environment. New York: Academic Press; 1981.
- [Background] Bernstein DP, Fink L. Childhood Trauma Questionnaire: A retrospective self-report manual. San Antonio, Texas: The Psychological Corporation; 1998.
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. J Psychopathol Behav Assess. 2016 Sep;38(3):443-55.
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difﬁculties in Emotion Regulation Scale. J Psychopathol Behav Assess. 2003;15.
- [Background] Gross JJ. The emerging field of emotion regulation: An integrative review. Rev Gen Psychol. 1998;2(3):271-99.
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Meunier D, Lambiotte R, Fornito A, Ersche KD, Bullmore ET. Hierarchical modularity in human brain functional networks. Front Neuroinform. 2009 Oct 30;3:37. doi: 10.3389/neuro.11.037.2009. eCollection 2009. PMID 19949480
- [Background] Nolte J. The human brain: an introduction to its functional anatomy. 4th ed. St. Louis, MO: Mosby; 2008.
- [Background] Rusted J, Sheppard L, Waller D. A Multi-centre Randomized Control Group Trial on the Use of Art Therapy for Older People with Dementia. Group Anal. 2006 Dec 1;39(4):517-36.
- [Derived] Wu-Chung EL, Bonomo ME, Brandt AK, Denny BT, Karmonik C, Frazier JT, Blench K, Fagundes CP. Music-induced cognitive change and whole-brain network flexibility: a pilot study. Front Neurosci. 2025 Jun 5;19:1567605. doi: 10.3389/fnins.2025.1567605. eCollection 2025. PMID 40538861
- See also: The Rice Arts, Cognition, and Health Science Initiative website. — http://arches.rice.edu/